## **Consent for Photography**

Title: A Randomized Controlled Trial on the Application of Artificial Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical Care Nurses

NCT Number: Not Available as yet

Document Date
December 5, 2025

## مستشفى الملك فيصل التخصصي ومركز الابحاث

## KING FAISAL SPECIALIST HOSPITAL AND RESEARCH CENTRE

| USE ONLY | | |
|---|---|---|
| I hereby authorize the Hospital Authorized Personnel to photograph<br>me and/or take electronic records of me for one or more of the<br>following reasons:<br>( Delete if inapplicable ) | | بهــذا أفوض موظفي المس<br>تسجيلات الكترونية للسبب<br>(اشطب البند الذي لاينطيق) |
| <ul> <li>1 - Medical Records</li> <li>2 - Publication in a medical journal</li> <li>3 - Medical Teaching</li> <li>4 - Other (Please specify)</li> </ul> | خدیدها) | <ol> <li>للسجلات الطبية</li> <li>للنشر في المجلة الطبية</li> <li>للتعليم الطبي</li> <li>لأسباب أخرى (يرجى ألم</li> </ol> |
| I understand that my refusal to sign this consent would not change the course of my treatment. | وقيع على هذا الاذن الخطي لن يؤثر على سير | أعلم أن احجامي عن التر<br>معالجتي. |
| I voluntarily consent to this procedure and hereby release King Faisal Specialist Hospital and Research Centre, the Physicians and other personnel working with the institution from any legal liability associated with this procedure. | لاجراء فانني أعفي مستشفى الملك فيصس<br>ث والأطباء والموظفين العاملين فيه من أي<br>م هذا الاجتراء . | وبمسوافقتي على هذا اأ<br>التخصصي ومركز الأبحساء<br>مسئوليات قانونية تترتب علم |
| Printed Names and Signatures | هاء مكتوبة بوضوح والتوفيعات<br>، | الأسي |
| Witness الثنامد | Patient | المريض |
| Physician الطبيب | Date | التاريخ |
| In case the patient's condition reasonably precludes the ability to grant informed consent, the above information has been explained to the following responsible relative and treatment is hereby authorized. | سمح بمنح هذا الأذن الموافقة فانه قد تـم<br>(ه الـي ولـي الأمر والـذي وافـق علـي التوقيـه | نظـرا لأن حالـة المـريـض لاتـ<br>شـرح المعلومـات الـواردة اعــلا |
| In case the patient's condition reasonably precludes the ability to grant informed consent, the above information has been explained to the following responsible relative and treatment is hereby au- | سمح بمنح هذا الأذن الموافقة فانه قد تـم<br>(ه الـي ولـي الأمر والـذي وافـق علـي التوقيـه | |

| octor's Instructions: | تعليهات الأطباء |
|---|---|
| BODY PART AP PA LAT 3/4 CLOSE UP UP | ALL PHOTOGRAPHS ARE THE PROPERTY OF KFSH & RC |
| (Important : Please include for retrieval purpose) OPIES TO : | |